CLINICAL TRIAL: NCT00112749
Title: Does Blocking Proinflammatory Cytokines Diminish Cancer-Related Fatigue?
Brief Title: Infliximab in Treating Cancer-Related Fatigue in Postmenopausal Women Who Have Undergone Treatment for Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment stopped due to slow accrual and lack of evidence of need for further continuation of protocol in inpatient setting.
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000428460; UCLA-0410033-01
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2016-02

CONDITIONS: Breast Cancer; Fatigue
Keywords: stage I breast cancer; stage II breast cancer; breast cancer in situ; fatigue
MeSH Terms: conditions — Breast Neoplasms; Fatigue; Breast Carcinoma In Situ | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study Arm (Experimental): Please see intervention description
  Interventions: Biological: infliximab; Other: Clinical Assessment; Other: Self-report questionnaires; Other: Immune Assessment

INTERVENTIONS:
Biological: infliximab — A single infusion of 1mg/kg will be administered.
Other: Clinical Assessment — Medical, psychiatric, and immune evaluation.
Other: Self-report questionnaires — Fatigue Symptom Inventory, Multidimensional Fatigue Symptom Inventory, Hamilton Depression Rating Scale, Beck Depression Inventory II, Hamilton anxiety Rating Scale, Pittsburgh Sleep Quality Index, Brief Pain Inventory, MOS SF-36.
Other: Immune Assessment — Proinflammatory cytokines and markers of cytokine activity and lymphocyte subsets and CBC.

SUMMARY:
RATIONALE: Infliximab may help improve energy levels in patients who have undergone treatment for breast cancer.

PURPOSE: This phase II trial is studying how well infliximab works in treating cancer-related fatigue in postmenopausal women who have undergone treatment for stage 0, stage I, or stage II breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the association between the body's immune system and energy, sleep, mood, and other symptoms in postmenopausal women who have undergone treatment for stage 0-II breast cancer.
* Determine whether treatment with infliximab affects energy and immune function in these patients.

OUTLINE: Patients receive infliximab IV over 2 hours.

Patients complete a diary twice daily for 14 days before and for 14 days after infliximab administration to assess fatigue and other symptoms, including mood, pain, and sleep.

After completion of study treatment, patients are followed at 2 weeks and then monthly for 3 months.

PROJECTED ACCRUAL: A total of 10 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Women who report elevated fatigue following cancer diagnosis and treatment

Exclusion Criteria:

* Women who have medical conditions that may affect the immune system or are associated with baseline fatigue syndrome, and/or who use medications that affect the immune system or fatigue.
* Women with major affective disorders and those with sleep or pain disorders.
* Presence of medical conditions that may but subject at undue risk for experimental procedures.
* Chronic or recurring infections, symptoms of chronic heart failure, demyelinating disorders, and those taking immunosuppressive medications.
* Neoplastic disease other than primary breast cancer
* Compromised cardiovascular function
* Insulin-dependent diabetes
* Neurological disorder
* Peripheral neuropathy
* Pregnancy
* Use of psychotropic medications within 2 weeks of screening
* Abnormal screening laboratory findings (i.e., creatinine > 1.4mg%; anemia; abnormal thyroid hormone; hematuria; elevated liver function tests, low protein or albumin; fasting glucose >120mg%; elevated FTI or TSH; positive TB screening, HIV screening or hepatitis C).
* Smokers

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2005-02; Primary Completion 2007-01 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Change in fatigue as measured by the fatigue symptom inventory (FSI) | At baseline and after completion of study treatment, 4 years
Change in fatigue as measured by multidimensional fatigue symptom inventory (MFSI) | At baseline and after completion of study treatment, 4 years

SECONDARY OUTCOMES:
Change in proinflammatory cytokines as measured by interleukin-1 receptor antagonist value | At baseline and after completion of study treatment, 4 years
Change in proinflammatory cytokines as measured by interleukin 6 value | At baseline and after completion of study treatment, 4 years
Change in proinflammatory cytokines as measured by tumor necrosis factor | At baseline and after completion of study treatment, 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Patricia A. Ganz, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States